CLINICAL TRIAL: NCT06161168
Title: Bootle Blast, a Movement Tracking Video Game for Home-based Motor Therapy: Understanding the Family Experience
Brief Title: Bootle Blast: Understanding the Family Experience
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 0110
Record Dates: First submitted 2023-07-25; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-08

CONDITIONS: Cerebral Palsy; Developmental Coordination Disorder; Developmental Disability; Autism Spectrum Disorder; Spinal Cord Injuries; Stroke; Acquired Brain Injury; Motor Skills Disorders
Keywords: Hand function; Arm function; At-home rehabilitation; Trunk stability; Balance
MeSH Terms: conditions — Cerebral Palsy; Motor Skills Disorders; Developmental Disabilities; Autism Spectrum Disorder; Spinal Cord Injuries; Stroke; Brain Injuries

STUDY DESIGN:
Intervention Model Description: This is a 17 week mixed methods study with a non-blinded, randomized, multiple baseline single-case experimental design (SCED) to answer the secondary research question. The research design has two phases: a baseline phase (A) wherein a representative baseline will be established through repeated measurements of the PQRS, followed by the Bootle Blast intervention phase (B). In a randomized, multiple baseline SCED, the start of the B phase is randomized to mitigate threats to internal validity. A minimum of 3 measurements is required in each phase. In this study, participants will be randomly allocated to a baseline A phase ranging from 10 to 21 days. The B Phase will be 8 weeks followed by a second 3 week A phase. Families will retain Bootle Blast at home and will have the option to continue use of Bootle Blast in weeks 15 to 17 as desired.
Masking Description: Assessors will be trained on practice videos prior to establish consistent scoring practices. Additionally, assessors will be blinded to the time point at which the video recording was collected. Lastly, blinded therapists will observe gameplay videos collected at the beginning and towards the end of the intervention to identify movements made, any compensatory movements observed, repetition counts, fatigue level, as well the child's overall coordination (i.e. the smooth and controlled use of movements in motor performance with consideration of timing, velocity, targeting accuracy, motor planning, directions, force and endurance).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Baseline Phase (10 or 21 days) (Experimental): In this study, participants will be randomly allocated to a baseline (A) phase that is further divided into two sub-phases, with different durations of either 10 or 21 days. The allocation to different durations of the baseline phase is randomized in order to mitigate threats to internal validity. During the baseline (A) phase, a representative baseline will be established through repeated measurements of the PQRS. Following the baseline phase (A), the 8-week intervention phase (B) is implemented, followed by a second 3-week (A) phase. There is no separate control group in this study, and all participants receive the same intervention during the intervention phase (B).
  Interventions: Device: Bootle Blast Play Phase (B)

INTERVENTIONS:
Device: Bootle Blast Play Phase (B) — Bootle Blast will be trialed for 14 weeks in the homes of 60 young people (6 to 17 years) with any motor condition that could be addressed by the Bootle Blast system, regardless of their diagnosis. The investigators will assess feasibility (e.g. independent home setup, ability to set/meet self-directed play time goals), enablers/barriers to use, and perceived value.
  During the 8-week intervention phase (B), children will have Bootle Blast at home and play it according to their family-directed playtime goals. Weekly logs of therapy activities and problems encountered while playing will be collected through survey links. Additionally, families will record a video of their child performing the tasks associated with their COPM goals on a weekly basis. After the 8-week intervention (B) phase, participants will enter a second 3-week baseline (A) phase, during which they'll be asked to stop playing Bootle Blast, and the game will be programmatically locked to prevent further play.

SUMMARY:
One in 60 children have a physical disability that can impact activities and participation. Occupational and physical therapies can be of great benefit, but are costly and difficult to access. Working with children, parents and clinicians, the investigators developed a mixed reality video game, Bootle Blast, which children can play to develop motor skills. Using a 3D sensor, Bootle Blast tracks movements and manipulation of real-life objects. Since 2017, Bootle Blast has been used in clinics by Holland Bloorview, Canada's largest children's rehabilitation hospital. Home use of Bootle Blast has resulted in positive clinical outcomes for children with cerebral palsy. Bootle Blast is not yet commercially available and has yet to be trialed in "real-world" contexts.

To understand real-world implementation, Bootle Blast will be trialed for 14 weeks in the homes of 60 young people (6 to 17 years) with any motor condition that could be addressed by the Bootle Blast system, regardless of their diagnosis. The investigators will assess feasibility (e.g. independent home setup, ability to set/meet self-directed play time goals), enablers/barriers to use, and perceived value. User experience will inform product, training and resource development. The research team combines expertise in engineering design, medicine, physiotherapy, qualitative methods, commercialization, knowledge translation, and includes young people with lived experience.

DETAILED DESCRIPTION:
One in 60 Canadian children has a physical disability that impacts function, activity and participation. Physical and occupational therapies are important for improving/maintaining their coordination, flexibility, strength, dexterity and function. These therapies can enhance children's independence, education and employment opportunities, as well as leisure play and social inclusion. Therapies can also mitigate need for surgical intervention, secondary injuries and other complications that result from compensatory movements and poor conditioning as the child grows. While the benefits of therapy are significant, costs for families and the healthcare system are escalating. Demand for therapy outpaces availability. Families in rural areas may travel long distances to access services or miss out. Even when resources are available, therapy is seldom offered more than 1 or 2 times/week for 30 - 60 minutes while the literature suggests that 30 - 45 min of practice per day is necessary to drive neuroplastic change and motor learning. This underlies the need for home-based programs to increase opportunities for practice of goal-directed movements. While home-based therapy improves outcomes, nearly half of families report poor adherence due to limited time, lack of motivation, or forgetfulness. For parents, the role of "therapist at home" is associated with many challenges (i.e. structuring practices, ensuring good form, initiating/sustaining participation) and, in fact, can negatively impact parent-child relationships and elevate parental stress and burden of care. Maintaining child and parent motivation in home-based therapies is a long-standing challenge of great importance in pediatric practice. In fact, clinicians rate child motivation to be the most influential trait predicting success in motor therapies.

Movement-tracking video games for home-based therapy practice (i.e. therapy gaming) appeal to clinicians, children and parents. Video games are a popular pastime for 82% of children with disabilities and 88% of children without, with an average play time of 13 hrs/week. As such, therapy gaming is well aligned with the practice of family-centred care which favours treatments preferred by children.Therapy gaming is also compelling from a motor learning perspective with potential for intense practice, feedback, individualized programs, task specificity (i.e. similarity between virtual and real-world tasks), and social equalization. These five features are considered the "active ingredients" (i.e. reasons why a treatment is expected to be effective) of video games for motor therapy.

8 years ago, families and clinicians at Canada's largest children rehabilitation hospital, Holland Bloorview Kids Rehabilitation Hospital (Holland Bloorview), and partner organizations affiliated with Empowered Kids Ontario (EKO), asked: Can video games be used to create fun, effective opportunities for motor practice for children with CP? Finding no suitable technologies to deliver the active ingredients for motor therapy, the investigators partnered with knowledge users (i.e. children with disabilities, siblings, caregivers, clinicians), interdisciplinary researchers, specialists (e.g. engineers, games designers) and with guidance from provincial networks (CP-NET) and external partners (Toronto Innovation Acceleration Partners (TIAP), formerly MaRS Innovation; Ubisoft), developed Bootle Blast. Bootle Blast overcomes many established limitations of video games for motor therapy including: inability to target fine motor skills, solo gameplay and failure to sustain engagement without significant parent/therapist involvement. Bootle Blast is the first video game for motor therapy to apply best practices in motor learning, game design, and motivation theory. It provides high quality biofeedback and is built on a theoretical framework of engagement used in pediatric rehabilitation, as summarized in two systematic reviews the investigators generated in the research process. Using computer vision, Bootle Blast provides real-time feedback on skeletal movements and interactions with real-life objects used in gameplay (e.g. building blocks). This "mixed reality" play experience offers greater task specificity to enhance transfer of skills to everyday activities. It enables individualized treatment plans by supporting a wide range of motor skills with activities that can be calibrated to each child's abilities. Bootle Blast enables differently abled people to play together, enhancing social equalization.

Creating a product that can be successfully used at home by families as a complement to conventional therapies, as well as by those on waitlists or who no longer qualify for clinical services (e.g. children no longer considered for "early intervention"), will greatly expand the market potential of Bootle Blast.

OBJECTIVES. In this project, the investigators will conduct real-world testing to identify potential barriers to home use.

RESEARCH QUESTION: In this study, the investigators will answer the questions: Firstly, is it feasible for families to independently set-up and sustain use of Bootle Blast at home? And, secondly, does using Bootle Blast at home over 14 weeks impact perceived performance on family-identified goals? Bootle Blast will be considered feasible if: (i) >95% of families are able to setup Bootle Blast independently with assistance provided through online or telephone technical support if needed; and (ii) >70% of families achieve their self-identified playtime goal. The play time goal will be self-directed and inputted as part of the onboarding process. Adherence averages 70% in previous research. To answer the primary research question regarding feasibility for in-home implementation, the investigators will use mixed methods to explore challenges encountered in setting up and using Bootle Blast at home, its perceived value, and the enablers/barriers to engagement, including the types of supports desired by families. To answer the second research question regarding perceived impact, the investigators will use (i) the Canadian Occupational Performance Measure (COPM) to investigate changes in perceived performance on a family-identified primary goal associated with the Bootle Blast play and, (ii) the Performance Quality Rating Scale (PQRS). Survey and interview data will be used to provide further context. Finally, the investigators will conduct exploratory analyses into the accuracy of system-collected joint data and its potential to inform families/clinicians on changes in movement characteristics (e.g. smoothness of movement, reach envelope). The latter could provide families using the system at home with potentially useful information for progress tracking.

ELIGIBILITY:
Child Participant Inclusion Criteria:

* Any motor condition that can be addressed by the Bootle Blast system;
* Interest in developing motor skills practiced in BootleBlast;
* Aged 6-17 years;
* Sufficient cognitive capacity to play BootleBlast as indicated by caregiver/self report;
* Able to communicate in English;
* Intermittent access to internet;
* Ability to participate in video calling;
* Have a device to record and upload short videos;
* Have a caregiver willing to participate.

Child Participant Exclusion Criteria:

* Uncontrolled epilepsy triggered by video games;
* Medical condition making the physical activity in BootleBlast unsafe;
* Visual and/or hearing limitations affecting BootleBlast play;
* No access to internet at home
* Has previously participated in a study related to Bootle Blast.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-07-07 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | First and last day of Baseline Phase; 8th week of Intervention Phase; 3rd week of Follow-up Phase
  The family will complete the Canadian Occupational Performance Measure with the interviewer to establish 1 to 3 goals related to activities of everyday living (e.g. self-care, leisure) that they hope Bootle Blast might help with. The COPM assesses self-perceived performance and satisfaction on activities of importance to child/family. Participants then rate their performance and satisfaction for each goal/challenge area on a scale from 1 to 10 (low to high). Average scores for performance and satisfaction are calculated across the goals. The COPM is extensively used with children with CP in the target age range and with success in the research team's pilot work. It has good validity, responsiveness, reliability, and ability to track change over time. A change of 2 points on either the performance or satisfaction scale is considered clinically significant. The COPM takes ~20 minutes.
Performance Quality Rating Scale (PQRS) | Weekly throughout study completion (14 weeks)
  The PQRS will be used to evaluate parent-recorded videos of children performing one of their COPM each week. The PQRS is an observational, video-based tool that looks at actual performance on client-selected activities, and has been used in the context of SCED research for children with diverse diagnoses, including CP and DCD. It utilizes a 10 point scale with a score of 1 indicating ''can't do the skill at all'' and 10 indicating ''does the skill very well''. Quality takes into account, as applicable to the task, timeliness, accuracy, safety, and overall quality of performance or product. Ratings are based on average of completeness and quality. Inter-rater reliability for the PQRS is moderate ranging from 0.71-0.77. Test-retest reliability is also substantial (>0.9) across time periods and multiple raters. Assessors will be trained on practice videos to establish consistent scoring practices. Assessors will be blinded to the time point at which the video recording was collected.

SECONDARY OUTCOMES:
Rates of recruitment and attrition | Throughout study (17 weeks)
  This will inform the appropriateness of Bootle Blast to meet family's needs (e.g. interest in the system, availability of an appropriate space etc.). Reasons for non-participation will be recorded where possible.
Family Information Demographic Form | Following consent but prior to commencement of baseline phase (i.e. Week 0)
  The investigators will document demographic data on participants (e.g. gender, age, diagnosis), family (e.g. family composition, socioeconomic status, access to services) and the caregiver (e.g. comfort with technology, relationship with child), including relevant functional assessments (e.g. MACS and GMFCS level for CP; Movement ABC Battery61 for DCD) for descriptive purposes and to provide context for data synthesis. This survey will be hosted on REDcap and distributed via email links prior to the pre-intervention interview with a a maximum 3 reminders to ensure questionnaire completion. Any missing data or participant questions will be reviewed in the pre-intervention interview.
The ABILHAND-Kids | Week 0; 8th week of Intervention Phase; 3rd week of Follow-up Phase
  This will be used to describe the population in terms of level of functional ability and as an outcome measure. This questionnaire asks parents to report on their child's ability to perform 21 primarily bimanual activities on a 3 point scale (0=impossible, 1=difficult, 2=easy). The total maximum score is 42. Previous work has established its excellent test-retest reliability, inter-rater reliability, and internal consistency when completed by parents for children with CP aged 4 to 18 years. The 10 min survey has demonstrated sensitivity to change with a large effect size of 0.92 (logit change of 1.06) reported for children with CP aged 6-12 years and a moderate effect size (logit change of 0.71) for 13-19 year olds after treatments. Additionally, this questionnaire has good psychometric properties and use in a range of developmental conditions as may be included in this study. This parent-reported survey will be administered via REDCap.
The Pediatric Evaluation of Disability Inventory Computer Adaptive Test (PEDI-CAT) | Day 1 of Baseline Phase; 8th week of Intervention Phase; 3rd week of Follow-up Phase
  This is a participant-reported measure of functional skills in four domains, including performance of activities of daily living, mobility, social-cognitive, and responsibility. It has been used to both quantify function and measure change following interventions. It has strong validity and reliability in diverse populations with developmental disabilities across multiple age ranges. The online questionnaire will be filled out during the pre-intervention interview via screen share with the researcher reading the questions as needed and the participant indicating their responses. The assessment takes about 12 minutes.
Children & Adolescent Scale of Participation (CASP) | Week 0; 8th week of Intervention Phase; 3rd week of Follow-up Phase
  The CASP consists of 20 ordinal-scaled items and four subsections: 1) Home Participation (6 items), 2) Community Participation (4 items), 3) School Participation (5 items), and 4) Home and Community Living Activities (5 items). The 20 items are rated on a four-point scale: "Age Expected (Full participation)," "Somewhat Restricted," "Very Restricted," "Unable." It can be used with children 5 years and up. The CASP has excellent test re-test reliability (Intraclass Correlation Coefficient = 0.94), internal consistency (α ≥ 0.96) and construct and discriminant validity. The CASP will be completed by parents and by youth (>11 years) as previous research indicates that there may be differences between parent and youth reported participation. The CASP will be administered via REDCap.
Pre-intervention interview | Day 1 of Baseline Phase
  A 1 hour zoom interview will be conducted to understand each families' hopes/expectations for the Bootle Blast program and to establish the COPM goals (described below), one of which must be an activity conducive to weekly filming. During this interview, parents will be trained on how to record a video of their child performing the activity associated with one of their COPM goals and upload videos to Sync a secure cloud server (www.sync.com), as well as establish a consistent way of filming (e.g. appropriate lighting, consistent angle). To this end, the investigators will provide families with a tripod as needed to facilitate filming and may make suggestions such as marking the position where the tripod should be placed with a piece of tape, etc. This video will be used to complete the Performance Quality Rating Scale (PQRS), as described below.
Observation of the device set-up: Time Required | Last day of Baseline Phase
  Observations of the home set-up will be logged by researchers observing by video call using the observation checklist. The researcher will take note of the total time taken by participants to set up the Bootle Blast from start to finish (minutes). The home set up session will be recorded via the Zoom platform.
Observation of the device set-up: User Manual Utilization | Last day of Baseline Phase
  Observations of the home set-up will be logged by researchers observing by video call using the observation checklist. The researcher will take note of the frequency and duration of user manual consultation during the setup process (minutes). The home set up session will be recorded via the Zoom platform.
Observation of the device set-up: Complexity of Bootle Blast Setup Process | Last day of Baseline Phase
  Observations of the home set-up will be logged by researchers observing by video call using the observation checklist. The researcher will take note of the main points of confusion and number of errors made during the setup as noted by the observer through qualitative descriptions. The home set up session will be recorded via the Zoom platform.
Observation of the device set-up: Participant Interaction with Setup Components | Last day of Baseline Phase
  Observations of the home set-up will be logged by researchers observing by video call using the observation checklist. The researcher will take note of the the process of installing the Orbbec, setting up the game space, launching the game, and the involvement of children/caregivers during the setup through qualitative descriptions and Installation Success Rate (binary: yes/no). The home set up session will be recorded via the Zoom platform.
Observation of the device set-up: Onboarding Effectiveness | Last day of Baseline Phase
  Observations of the home set-up will be logged by researchers observing by video call using the observation checklist. The researcher will take note of how users interact with the game guide, calibration, playtime goal setup, game navigation, playing a mini-game through qualitative descriptions and Calibration Success Rate (binary: yes/no). The home set up session will be recorded via the Zoom platform.
Observation of the device set-up: Affective Responses | Last day of Baseline Phase
  Observations of the home set-up will be logged by researchers observing by video call using the observation checklist. The researcher will take note of the emotional responses of participants during the installation process through qualitative descriptions. The home set up session will be recorded via the Zoom platform.
System collected data | Throughout intervention phase (Week 1 - 8); Optional Phase (Week 15 - 17)
  All user activity (e.g. games played, time, skeletal joint movement data etc.) is recorded. Active (e.g. therapeutic movement) and passive (e.g. navigating menus) play time and the number of intentional therapeutic movements will be recorded. Periodically, the game will ask the player if they are having fun, if the challenge level is right, and if they are feeling tired. Video recordings collected via Bootle Blast are mostly non-identifying. The face and much of the background, are blocked to preserve privacy. Families can enable or disable video recordings which they can adjust at any time. Data will be encrypted, uploaded, and stored on Google Cloud's Firebase Realtime Database and Cloud Storage (Montreal-based server). Data are linked to the participant via a unique ID. No personal health information is collected or stored on the server. Upon study completion, participant data are removed from Google Cloud and transferred to a secure server located onsite at Holland Bloorview.
Child and Adolescent Factors Inventory (CAFI) | Following consent but prior to commencement of baseline phase (i.e. Week 0)
  The family will complete the CAFI to describe their child's challenges and strengths. This survey will be hosted on REDcap and distributed via email links prior to the pre-intervention interview with a a maximum 3 reminders to ensure questionnaire completion. Any missing data or participant questions will be reviewed in the pre-intervention interview.
Access To Therapy Services Questionnaire | Following consent but prior to commencement of baseline phase (i.e. Week 0)
  The family will complete the Access to Therapy Services questionnaire to describe their child's access to care and utilization of healthcare services. This survey will be hosted on REDcap and distributed via email links prior to the pre-intervention interview with a a maximum 3 reminders to ensure questionnaire completion. Any missing data or participant questions will be reviewed in the pre-intervention interview.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Biddiss, PhD, Principal Investigator — Bloorview Research Institute
Locations (1):
- Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No